CLINICAL TRIAL: NCT05579223
Title: Intrathecal Hydromorphone for Postoperative Pain of Anorectal Surgery: A Randomized, Double-blind, Parallel, Placebo-controlled Trial
Brief Title: Intrathecal Hydromorphone for Postoperative Pain of Anorectal Surgery
Acronym: IMPAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-22-005
Record Dates: First submitted 2022-09-28; First posted 2022-10-13 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-11

CONDITIONS: Acute Pain; Post Operative Pain; Anorectal Disorder; Analgesia
Keywords: hydromorphone; intrathecal opioid; post operative pain; anorectal surgery; placebo
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Rectal Diseases; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Hydromorphone Group (ITHM) (Experimental): Dosage Form: Hydromorphone Hydrochloride Injection 2mg:2ml. Dosage: 75 μg+ 5% glucose injection diluted to 1.5ml. Frequency and Duration: i.t., st
  Interventions: Drug: Intrathecal Hydromorphone Mono Injection
- Intrathecal Placebo Group (ITPO) (Placebo Comparator): Dosage Form: 5% glucose injection, 100ml/Package. Dosage: 1.5ml. Frequency and Duration: i.t., st
  Interventions: Drug: Intrathecal Placebo Mono Injection

INTERVENTIONS:
Drug: Intrathecal Hydromorphone Mono Injection — Experimental Drug: Hydromorphone Hydrochloride Injection. Administration: subarachnoid space mono bolus inject, + 5% glucose injection diluted to 75 μg:1.5ml, Speed ≤ 0.5 ml/s
  Other Names: ITHM
  Arms: Intrathecal Hydromorphone Group (ITHM)
Drug: Intrathecal Placebo Mono Injection — Placebo: 5% glucose injection. Administration: subarachnoid space mono bolus inject, 1.5ml, Speed ≤ 0.5 ml/s
  Other Names: ITPO
  Arms: Intrathecal Placebo Group (ITPO)

SUMMARY:
Anorectal problems, such as hemorrhoids, fistula, fissures, Etc., often require surgical treatment. Patients often have postoperative pain after these surgeries, which increases discomfort and hospital length of stay. The efficacy of oral non-opioids in the treatment of such pain is poor. Hydromorphone is an opioid analgesic commonly used orally or intravenously for postoperative pain management. We designed this trial to investigate the efficacy and safety of intrathecal (delivery directly to the spinal cord during spinal anesthesia) single dose hydromorphone versus intrathecal placebo in treating postoperative pain among human subjects after anorectal surgery, but also the recovery of postoperative motor capacity in these human subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical Diagnosis of anorectal disease, ready to undergo elective surgery
* 2. American Society of Anesthesiologists(ASA) physical status I-II
* 3. Desire to have a spinal anesthesia
* 4. Must be able to follow the medication dose and visit schedule

Exclusion Criteria:

* 1. Any contraindications to spinal anesthesia and intrathecal analgesia.
* 2. Complex co-morbidities, including

  1. Severe infection,
  2. Respiratory insufficiency,
  3. History of psychiatric or neurological disorders and other cognitive impairments
* 3. Chronic pain syndrome or current opioid use >10mg oral morphine equivalents/day
* 4. Allergy or intolerance to hydromorphone, NSAIDs and Cox-2 selective Inhibitor
* 5. Clinical diagnosis of obstructive sleep apnea syndrome(OSAS)
* 6. History of drug abuse
* 7. Women who are breastfeeding or pregnant
* 8. Participation in other clinical trials within three months
* 9. Already participated in this study once
* 10. Not considered suitable for the clinical trial by the investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale Pain Scores (NRS score for pain) | Time of spinal injection finished will be noted as time: "0". NRS, with movement 12 hours, will be collected by patient interview at 12 hours after spinal administration.
  NRS for pain (0-10) with movement 12 hours after spinal administration

SECONDARY OUTCOMES:
NRS score at rest/with movement | Time of spinal injection finished will be noted as time: "0". NRS, with movement or at rest, will be collected by patient interview at 1, 3, 6, 12, 24 and 36 hours after spinal administration.
  NRS score for pain (0-10) with movement, and at rest.
Highest pain NRS (0-10) in previous 12 hours | At 12 hours after spinal administration.
  NRS score for pain (0-10) with movement or at rest and the time.
Severity and incidence of any opioid-related complication at each time point | All data will be collected by patient interview at 1, 3, 6, 12, 24 and 36 hours after spinal administration.
  Including: nausea, vomiting, constipation, diarrhea, itching, dry mouth, dizziness, numbness, depression, anxiety, fever, skin rash, urinary retention, Etc.
Total non-opioid analgesic consumption | All data will be collected by patient interview at 12, 24 and 36 hours after spinal administration.
  Total non-opioid analgesic consumption at 12, 24 and 36 hours after spinal administration, mainly intravenous parecoxib/ketorolac/flurbiprofen injection dosage.
Recovery of lower extremity strength. | Data will be collected by patient interview at 12 hours after spinal administration.
  Time required to the recovery of casual movement of the lower extremities
Quality of Recovery Scale (QoR) | At 12, 24 and 36 hours post spinal administration.
  40-item quality of recovery score, QoR-40

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Xu, M.D., Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
This trial's study protocol, case report forms, Etc., is written in Chinese as the primary language. The Ethics Committee and the Human Genetic Resources Office have approved this trial. After completing the last follow-up, we will upload the translated versions as soon as possible.